CLINICAL TRIAL: NCT04678063
Title: Validation Study of the ALYATEC Allergen Exposure Chamber (EEC) by Determining the Concentration of Cat Allergen Inducing Early and/or Late Bronchial Response in Asthmatic Subjects Allergic to Cat
Brief Title: Validation of Strasbourg Environmental Exposure Chamber ALYATEC in Cat Allergic Subjects With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: ALY-003
Record Dates: First submitted 2020-12-04; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Allergic Asthma; Allergy; Allergy to Cats
Keywords: Cat allergy; Allergic rhinitis; Allergy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, cross-over study including two study groups
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthmatic subjects allergic to cat (Experimental): Group A will be randomized into 2 subgroups of 10 subjects: group A1 and A2. Both subgroupes will be exposed to placebo on exposure 1 then Subgroup A1 will be exposed to dose A on exposure 2 and dose B on exposure 3. Subgroup A2 will be exposed to dose B on exposure 2 and dose A on exposure 3. Dose A and B correspond to different Allergen concentration in the EEC.
  Interventions: Other: Exposure to Placebo; Other: Exposure to dose A and dose B of cat allergen
- Asthmatic allergic subjects not sensitized to cat (Active Comparator): Group B will be exposed to placebo at exposure 1, and then at exposure 2, the concentration of cat allergens corresponding to the dose that achieved the main objective (Dose A or B).
  Interventions: Other: Exposure to Placebo; Other: Exposure to a single dose of cat allergen

INTERVENTIONS:
Other: Exposure to Placebo — Patients are exposed to placebo in the EEC
Other: Exposure to dose A and dose B of cat allergen — Patients are exposed to dose A and B for successive exposures in the EEC
  Arms: Asthmatic subjects allergic to cat
Other: Exposure to a single dose of cat allergen — Patients are exposed to a single dose of cat allergen in the EEC according to the dose selected to achieve the main objective (dose A or B)
  Arms: Asthmatic allergic subjects not sensitized to cat

SUMMARY:
This is a randomized, double blind, cross-over study designed to determine the concentration of airborne cat allergen inducing bronchial response in asthmatic subjects allergic to cat, during allergen exposures in the Alyatec environmental exposure chamber (EEC).

The study was also designed to validate the specificity of the asthmatic reaction induced by exposure to airborne cat allergen in Alyatec EEC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having signed the informed consent
* Subjects affiliated to a social security scheme
* Non-specific bronchial hyperreactivity (HRBNS) assessed by a positive methacholine test
* FEV1 value > 70% of theoretical FEV1 value
* Asthma Control Test (ACT) ≥ 20/25 in 4 weeks prior to EEC exposure
* Women of childbearing potential should have a negative pregnancy test throughout the study period with effective contraception.

Group A:

* Cat allergic asthma (GINA 1, 2) associated with rhinitis and / or conjunctivitis symptoms triggered during an exposure to a cat.
* Positive skin prick-test to cat allergen extract (wheal diameter >3 mm compared to the negative control) Specific immunoglobulin E (IgE) for cat allergen > 0.7 kU/L

Group B:

* Mild allergic asthma (GINA 1 or 2) not sensitized to cat allergen with associated rhinitis and/or conjunctivitis.
* Negative skin prick-test and specific IgE for cat allergen
* Positive skin prick-test and specific IgE for another allergen.

Exclusion Criteria:

* Uncontrolled asthma, ACT asthma control questionnaire less than 20, in the last 4 weeks
* Uncontrolled asthma 2 weeks after interruption of LABA
* Long-term treatment by LABA, within 2 weeks prior to inclusion
* Existence of a severe obstructive syndrome with FEV1 <70% of the theoretical value
* Obstruction triggered by spirometric evaluations
* Hospitalization for asthma or exacerbation in the last 4 weeks
* Subjects treated with oral corticosteroids in the 4 weeks prior to inclusion in the study
* History of severe acute asthma requiring hospitalization in intensive care or intubation
* Subjects treated with biotherapy in the 4 months prior to inclusion in the study
* Presence of a cat at home, or daily exposure to cat allergens
* Desensitization to cat allergens in the last 6 months
* Active tobacco: plus 10 cigarettes / day or tobacco history plus 10 PA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
Determine the concentration of cat allergen (in ng/m3 of Der p1) necessary to induce a bronchial response in at least 60% of asthmatic subjects allergic to cat. | 10 hours: 4 hours of exposure in EEC then 6 hours post-exposure
  The bronchial response is evaluated by measuring FEV1 value.
  Early asthmatic response (EAR) occurs when a 20 percent drop in FEV1 is detected during the exposure compared to the pre-exposure FEV1.
  Late bronchial response (LAR) occurs when a 15 percent drop in FEV1 or 20 percent drop in peak flow is detected 1 to 6h after the EAR.

SECONDARY OUTCOMES:
Evaluate the safety of allergenic exposure in EEC | 28 hours: 4 hours of exposure in EEC then 24 hours post-exposure
  Safety is assessed with an asthma symptom self-report questionnaire performed during the 4h exposure and for 24h after the end of the exposure.
  The score was obtained from the sum of all four individual symptom scores (chest tightness, cough, wheezing and dyspnea) with a total possible score ranging from 0 (no symptoms) to 16 (maximum symptom intensity).
Evaluate the allergen concentration in the EEC | 4 hours exposure in EEC
  The measurement of allergen concentration is performed with several sensors positioned in the chamber.
Evaluate the specificity of the bronchial response | 4 hours exposure in EEC
  The specificity of the bronchial response is assessed with the exposure to cat allergen in the EEC of asthmatic allergic subjects non sensitized to cat.
Evaluate the effect of the exposure on rhinitis symptoms | 28 hours: 4 hours of exposure in EEC then 24 hours post-exposure
  The effect of the exposure on the rhinitis response is assessed with Total Nasal Symptom Score (TNSS).
  The TNSS was obtained from the sum of all four individual symptom scores, with a total possible score ranging from 0 (no symptoms) to 12 (maximum symptom intensity).
Evaluate the effect of the exposure on conjunctivitis symptoms | 28 hours: 4 hours of exposure in EEC then 24 hours post-exposure
  The effect of the exposure on the conjunctivitis response is assessed with Total Ocular Symptom Score (TOSS).
  The TOSS was obtained from the sum of all four individual symptom scores, with a total possible score ranging from 0 (no symptoms) to 12 (maximum symptom intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric de Blay, Pr., Principal Investigator — Alyatec
Locations (1):
- Alyatec, Strasbourg, Grand Est, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alyatec website — https://www.alyatec.com/en/